CLINICAL TRIAL: NCT06791772
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of CM313(SC) Injection in Subjects With Systemic Lupus Erythematosus
Brief Title: Study of CM313(SC) Injection in Systemic Lupus Erythematosus(SLE)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CM313-106106
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): CM313
  Interventions: Biological: CM313 injection
- Group B (Experimental): CM313
  Interventions: Biological: CM313 injection
- Group C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM313 injection — CM313 600mg（4ml）/vial. Subcutaneous injection 600mg. The first 5 doses were administered weekly, followed by every two weeks, a total of 14 doses.
  Arms: Group A
Biological: CM313 injection — CM313 600mg（4ml）/vial. Subcutaneous injection 1200mg. The first 5 doses were administered weekly, followed by every two weeks, a total of 14 doses.
  Arms: Group B
Drug: Placebo — Placebo 4 mL/vial. Subcutaneous injection 4 or 8 mL. The first 5 doses were administered weekly, followed by every two weeks, a total of 14 doses.
  Arms: Group C

SUMMARY:
To evaluate the efficacy and safety of CM313(SC) injection in systemic lupus erythematosus(SLE)

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 65 years.
2. Voluntarily signed the informed consent form (ICF).
3. Patients were diagnosed with systemic lupus erythematosus(SLE) according to the diagnostic classification criteria of the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) in 2019.
4. Systemic Lupus Erythematosus Disease Activity Index - 2000(SLEDAI-2K) score ≥6 during screening, and SLEDAI-2K clinical score (except for low complement and/or positive anti-dsDNA antibodies) ≥4 during screening and at baseline.
5. Positive antinuclear antibody and/or anti-dsDNA antibody results defined in accordance with the laboratory reference value range of the Central laboratory during the screening.
6. ≥1British Isles Lupus Assessment Group-2004 (BILAG-2004) organ system rated as A or ≥ 2 organ system rated as B, and Physician's Global Assessment(PGA) score ≥1.0 during screening.
7. Maintain a stable standard treatment regimen for at least 30 days prior to initial dosing of the investigational product.

Exclusion Criteria:

1. Kidney disease: Severe lupus nephritis within within 8 weeks prior to randomization.
2. Patients with systemic lupus erythematosus(SLE) or non-SLE related central nervous system disease within 8 weeks prior to randomization.
3. There were non-SLE inflammatory skin or joint diseases that the investigators thought might be evaluated during the screening period.
4. History of clinically significant diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving Systemic Lupus Erythematosus Responder Index -4 (SRI-4) | Up to week 24
  SRI-4 response is defined as:
  * Systemic Lupus Erythematosus Disease Activity Index - 2000 (SLEDAI-2K) reduction from baseline of ≥ 4 points
  * No British Isles Lupus Assessment Group-2004 (BILAG-2004) worsening, defined as ≥ 1 new A or ≥ 2 new B items compared to baseline
  * No worsening in Physician's Global Assessment (PGA), defined as an increase of ≥ 0.3 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China